CLINICAL TRIAL: NCT03849404
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Active Control Study to Compare the Efficacy, Safety, and Immunogenicity of AVT02 Versus Humira® in Patients With Moderate-to-Severe Chronic Plaque Psoriasis (ALVOPAD PS)
Brief Title: Efficacy, Safety, and Immunogenicity of AVT02 With Moderate-to-Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT02-GL-301
Record Dates: First submitted 2019-02-05; First posted 2019-02-21 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2019-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT02 100mg/mL (Adalimumab Biosimilar) (Experimental): Patients will be randomized to AVT02 on 1: 1 basis from the dosing day of Day 1 until week 48
  Interventions: Biological: Adalimumab
- EU-Humira 100mg/mL (Adalimumab Originator) (Experimental): Patients will be randomized to EU-Humira on 1: 1 basis from the dosing day of Day 1 until week 48
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Patients in AVT02 arm will receive an initial loading dose of AVT02 80 mg (2 × 40 mg) administered subcutaneously (SC), followed by 40 mg given SC once every other week (EOW) starting 1 week after the loading dose, and will continue to receive AVT02 until Week 48 Patients in EU-Humira arm will receive an initial loading dose of Humira 80 mg (2 × 40 mg) administered SC, followed by 40 mg given SC EOW starting 1 week after the loading dose and will continue to receive Humira until Week 48

SUMMARY:
Safety and Efficacy study of AVT02 (Alvotech Biosimilar to Adalimumab), in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
A Multicenter, Double-blind, Randomized, Parallel-group, Active Control Study to Compare the Efficacy, Safety, and Immunogenicity of AVT02 Versus Humira® in Patients with Moderate-to-Severe Chronic Plaque Psoriasis (ALVOPAD PS).

This study will be conducted at about 40 study centers in central and eastern European countries. A contract research organization, will oversee operational aspects of this study on behalf of Alvotech Swiss AG (Alvotech), the Sponsor of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate-to-severe chronic plaque psoriasis who has involved body surface area (BSA) ≥ 10% (Palm Method), ≥ 12 on the PASI, and static Physicians Global Assessments (sPGA) ≥ 3 (moderate) at Screening and at BL.
* Patient has had stable psoriatic disease for at least 2 months (ie, without significant changes as defined by the Investigator or designee).
* Patient is a candidate for systemic therapy and the patient has a previous failure, inadequate response, intolerance, or contraindication to at least 1 systemic antipsoriatic therapy including, but not limited to, methotrexate, cyclosporine, psoralen plus ultraviolet light A (PUVA), and ultraviolet light B (UVB).

Exclusion Criteria:

* Patient has prior use of 2 or more biologics for treatment of PsO.
* Patient diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (eg, eczema), or other systemic autoimmune disorder inflammatory disease at the time of the Screening visit that would interfere with evaluations of the effect of the study drug on psoriasis.
* Patient has prior use of any of the following medications within specified time periods or will require use during the study:

  1. Topical medications within 2 weeks of BL (Week 1).
  2. PUVA phototherapy and/or UVB phototherapy within 4 weeks prior to the BL Visit.
  3. Nonbiologic psoriasis systemic therapies (eg, cyclosporine, methotrexate, and acitretin) within 4 weeks prior to the BL Visit.
  4. Any prior or concomitant or biosimilar adalimumab therapy, either approved or investigational.
  5. Any systemic steroid in the 4 weeks prior to BL.

Note: Only key inclusion/exclusion criteria mentioned here. Patients will be screened and randomized per the list in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Baseline to Week 16
  Percent (%) change in Psoriasis Area and Severity Index (PASI)

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Percent improvement in PASI from BL to Week 8, 12, 24, 32, 42, and 50
  Percent (%) change in Psoriasis Area and Severity Index (PASI)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (20):
- Estonia (4):
  - Innomedica OU, Tallinn
  - OU Vahlberg & Pild, Tallinn
  - North Estonia Medical Centre Foundation, Dermatovenerology Centre, Tallinn
  - Tartu University Hospital, Dermatology Clinic, Tartu
- Georgia (5):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - The first University Clinic of Tbilisi State Medical University, Tbilisi
  - Scientific Research National Center of Dermatology and Venereology LLC, Tbilisi
  - Health Institute LLC, Tbilisi
  - David Abuladze Georgian-Italian Clinic LTD, Tbilisi
- Poland (10):
  - ClinicMed Daniluk, Nowak Spółka Jawna, Bialystok
  - NZOZ Osteo-Medic s.c. Artur Racewicz, Jerzy Supronik, Bialystok
  - Centrum Badań Klinicznych PI-House Sp. Z o.o., Gdansk
  - Synexus Polska Sp. z o.o. Oddział w Gdańsku, Gdansk
  - Center Med Kraków Sp. Z o.o., Krakow
  - Centrum Medyczna ALL-MED, Lodz
  - NZOZ "Nasz Lekarz" Sławomir Jeka, Praktyka Grupowa Lekarzy Rodzinnych z Przychodnią Specjalistyczną, Torun
  - Synexus Polska Sp. z o.o.Oddział w Warszawie, Warsaw
  - DermMedica Sp. z o.o., Wroclaw
  - Synexus Polska Sp. z o.o. Oddział we Wrocławiu, Wroclaw
- Zaporizhzhya Regional Dermatology and Venereology Clinical Dispensary, Zaporizhzhya, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feldman SR, Reznichenko N, Pulka G, Kingo K, George Galdava, Berti F, Sobierska J, Dias R, Guenzi E, Hendrik Otto, Haliduola HN, Kay R, Stroissnig H. Efficacy, Safety and Immunogenicity of AVT02 Versus Originator Adalimumab in Subjects with Moderate to Severe Chronic Plaque Psoriasis: A Multicentre, Double-Blind, Randomised, Parallel Group, Active Control, Phase III Study. BioDrugs. 2021 Nov;35(6):735-748. doi: 10.1007/s40259-021-00502-w. Epub 2021 Oct 16. PMID 34657274